CLINICAL TRIAL: NCT02893332
Title: Tyrosine-kinase Inhibitor （TKI） With or Without SBRT in Newly Diagnosed EGFRm Advanced Staged Lung Adenocarcinoma
Brief Title: Stereotactic Body Radiation Therapy (SBRT) in Newly Diagnosed Advanced Staged Lung Adenocarcinoma (Sindas)
Acronym: Sindas
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: After interim analysis, IRB recommend termination.
Sponsor: Sichuan Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, ming zeng, MD, Director of Cancer Center, Sichuan Provincial People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2016 15-1
Record Dates: First submitted 2016-08-24; First posted 2016-09-08 (Estimated); Last update posted 2021-02-03 (Actual); Status verified 2021-01

CONDITIONS: Stage IV EGFR Mutated Non-Small Cell Lung Cancer
MeSH Terms: interventions — Gefitinib; Erlotinib Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TKI without SBRT (Active Comparator): Newly diagnosed Patients will be placed on EGFR-TKI, ,Gefitinib 250mg po qd or Tarceva 150mg po qd for their metastatic EGFR-mutant stage IV oligometastatic disease.
  The oligometastatic disease will not receive SBRT
  Interventions: Drug: TKI (Gefitinib or Tarceva )
- TKI with SBRT (Experimental): experimental: Oligometastatic Non-Small Cell Lung Cancer Newly diagnosed patients will be placed on EGFR-TKI, Gefitinib 250mg po qd or Tarceva 150mg po qd, for their metastatic EGFR-mutant stage IV oligometastatic disease. All patients will TKI, Gefitinib 250mg po qd or Tarceva 150mg po qd, and SBRT at the same time.
  SBRT to up to 5 sites. The SBRT dose range from 5 Gy per fraction to 8 Gy per fraction. SBRT deliver within 5 fractions.
  Interventions: Radiation: Radiation: SBRT; Drug: TKI (Gefitinib or Tarceva )

INTERVENTIONS:
Radiation: Radiation: SBRT — A first line TKI (Gefitinib 250mg po qd or Tarceva 150mg po qd ) will be administered according to the standard dosing of the drug for metastatic NSCL during a 1-week run-in period after which SBRT will be delivered to the all oligometastatic lesions concurrently with the TKI. The SBRT dose will be , ranging from at 25Gy (5 Gy per fraction) to 40 Gy (8 Gy per fraction).
  Arms: TKI with SBRT
Drug: TKI (Gefitinib or Tarceva ) — A first line TKI (Gefitinib 250mg po qd or Tarceva 150mg po qd ) will be administered according to the standard dosing of the drug for metastatic NSCL, no local therapy apply to oligo-metastatic sites.

SUMMARY:
To tested if the adding of consolidative SBRT to TKI in EGFR mutated patients with less than or equal to 5 metastatic sites (primary + 5) will improve progression free survival (PFS) compared to TKI alone.

DETAILED DESCRIPTION:
This protocol is a randomized phase III trial of TKI versus consolidative Stereotactic Body Radiation Therapy (SBRT) plus TKI for patients with Stage IV non-small cell lung cancer (NSCLC).

Prior to accrual on the trial, patients with Stage IV NSCLC will be tested with positive EGFR mutation. Patients who with fewer than or equal to 5 sites of oligometastatic disease will be randomized toTKI or consolidative SBRT to all sites of disease (followed by TKI at the medical oncologist's discretion). Choices of TKI will be determined by the medical oncologist based on clinical appropriateness.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed metastatic lung adenocarcinoma (recurrent or de novo) harboring sensitizing EGFR mutations (L858R, exon 19 deletion, G719A, L861Q, S768I, exon 19 insertions) with oligometastatic disease (≤5 discrete lesions of disease irrespective of location, inclusive of the primary lesion):

  * all sites of disease must be amenable to definitive treatment with a local therapy (surgical resection, stereotactic radiosurgery, ablation and conventional radiation therapy) as determined by surgery, interventional radiology and radiation oncology
  * all intrathoracic lymph nodes (including hilar, mediastinal, and supraclavicular nodal disease) are considered 1 discrete lesion.
* No brain metastasis is allowed.
* Patients already started on erlotinib are eligible as long as their sites of disease are determined to be eligible for definitive local therapy by consensus of the principal investigators within 12 weeks of the patient first taking erlotinib.
* Lung adenocarcinoma histology confirmed
* Karnofsky Performance Status ≥ 70%
* Adequate bone marrow, liver and renal function, as specified below:

  * Absolute Neutrophil Count (ANC) ≥ 1.5 x 109/L
  * Hemoglobin ≥ 8 g/dL
  * Platelets ≥ 100 x 109/L
  * Serum total bilirubin ≤ 1.5 x upper limit of normal (ULN) (except for patients with documented Gilbert's Syndrome)
  * AST and ALT ≤ 2.5 x ULN or ≤ 5 x ULN if liver metastases are present
  * Serum creatinine ≤ 1.5 x upper limit of normal or creatinine clearance ≥ 60ml/min for patients with creatinine levels above institutional normal.
* For women of child-bearing potential, negative pregnancy test within 14 days prior to starting treatment
* Men and women of childbearing age must be willing to use effective contraception while on treatment and for at least 3 months thereafter

Exclusion Criteria:

* Treatment with TKI prior to developing metastatic disease
* Malignant pleural effusion or pleural disease
* Leptomeningeal disease or brain metastasis.
* Any site of disease that is not amenable to definitively local therapy including surgery or radiation therapy
* Women who are breastfeeding or pregnant
* Concurrent malignancies other than non-melanoma skin cancer that require active ongoing treatment.
* Any medical co-morbidities that would preclude surgery or radiation therapy

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2016-01-15 (Actual); Primary Completion 2020-08-30 (Actual); Study Completion 2020-08-30 (Actual)

PRIMARY OUTCOMES:
Progression free survival | 4 years
  Evaluate the effect of TKI with or without SBRT on progression free survival,to describe local control and out-of-field disease progression

SECONDARY OUTCOMES:
Overall survival | 4 years
  To evaluate overall survival after SBRT followed by maintenance chemotherapy in comparison to maintenance chemotherapy alone.
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability]) | 4 years
  Using CTCAE system to evaluate toxicity profile

CONTACTS AND LOCATIONS:
Overall Officials: Ming Zeng, MD PhD, Study Chair — Sichuan Provincial People Hospital
Locations (1):
- Sichuan PPH, Cancer Center, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Wang XS, Bai YF, Verma V, Yu RL, Tian W, Ao R, Deng Y, Zhu XQ, Liu H, Pan HX, Yang L, Bai HS, Luo X, Guo Y, Zhou MX, Sun YM, Zhang ZC, Li SM, Cheng X, Tan BX, Han LF, Liu YY, Zhang K, Zeng FX, Jia L, Hao XB, Wang YY, Feng G, Xie K, Lu Y, Zeng M. Randomized Trial of First-Line Tyrosine Kinase Inhibitor With or Without Radiotherapy for Synchronous Oligometastatic EGFR-Mutated Non-Small Cell Lung Cancer. J Natl Cancer Inst. 2023 Jun 8;115(6):742-748. doi: 10.1093/jnci/djac015. PMID 35094066